CLINICAL TRIAL: NCT01789710
Title: Contingency Management for Smoking Cessation in Homeless Smokers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Duke University (Other)
Collaborators: Durham VA Medical Center (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Pro00040194
Record Dates: First submitted 2013-02-08; First posted 2013-02-12 (Estimated); Last update posted 2015-06-12 (Estimated); Status verified 2015-06

CONDITIONS: Smoking; Homeless Persons
Keywords: smoking; homelessness; contingency management
MeSH Terms: conditions — Smoking | interventions — Bupropion; Nicotine Replacement Therapy; Nicotine; Tobacco Use Cessation Devices; Nicotine Chewing Gum

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Active Contingency Management (Experimental): All participants are assigned to a single arm, active contingency management. In this arm, participants are provided monetary rewards for remaining abstinent from smoking.
  Interventions: Drug: Bupropion; Drug: Nicotine replacement therapy; Behavioral: Contingency Management

INTERVENTIONS:
Drug: Bupropion — All participants who are medically eligible to take Bupropion will receive this study medication one week prior to their smoking quit date.
  Other Names: Zyban
Drug: Nicotine replacement therapy — All participants will receive two forms of nicotine replacement therapy - nicotine patches and a rescue method (either gum or lozenge).
  Other Names: Nicoderm CQ, Nicotine patch; Nicotine polacrilex, nicotine gum; Nicotine lozenge
Behavioral: Contingency Management — All participants will be asked to provide home carbon monoxide monitoring with equipment that is loaned to them. When participants provide readings that are low enough to suggest abstinence from smoking, they are provided monetary reinforcement (i.e., money).

SUMMARY:
The purpose of this study is to examine the effectiveness of an internet-based contingency management program for smoking cessation in persons who are homeless. Thirty homeless smokers will be enrolled in the study. Participants will receive payment based on their own low carbon monoxide readings, which indicate being quit from smoking. Participants will be prescribed nicotine replacement (patches and either gum or lozenge)and bupropion. All participants will receive a four sessions of smoking cessation counseling, and will be trained to perform carbon monoxide monitoring with a device provided by the study. They will also be provided with a mobile phone equipped with a video camera, and will use this equipment at home to monitor their carbon monoxide . Participants will record videos of themselves taking a carbon monoxide reading and displaying the results, and will upload the videos to a secured website that is only accessible by the research team members and the participant. Payment will be based on providing carbon monoxide readings that indicate abstinence.

The study is designed to address the following aims:

Specific Aim 1: To evaluate whether it is feasible to use internet-based contingency management for helping smokers who are homeless stop smoking.

Specific Aim 2: To evaluate how effective internet-based contingency managementis on decreasing smoking in smokers who are homeless.

ELIGIBILITY:
Inclusion Criteria:

* must be a Veteran who is eligible for care within the VA system;
* must be currently homeless or have been homeless more than twice in the past year period;
* must have current smoking status of at least 10 cigarettes per day for at least 1 year (verified with breath carbon monoxidemeasurement);
* must be aged 18 to 70;
* must be English speaker

Exclusion Criteria:

* Pregnancy;
* Any substance use disorder in any of the following drug categories: opioids, cocaine, alcohol, sedatives, stimulants, hallucinogens, or drugs categorized as "other" per the Structured Clinical Interview for Diagnostic and Statistical Manual-IV.
* Urine drug screen results positive for cocaine, amphetamines, stimulants, opioids, or hallucinogens;
* Not stable on medications for the study period;
* Use of any other forms of nicotine such as cigars, pipes, or chewing tobacco;
* Participants may be excluded if they have a seizure disorder, uncontrolled diabetes or an eating disorder;
* Prior history of hepatitis or cirrhosis; current hepatitis or cirrhosis
* Score less than 80 on Kaufman Brief Intelligence Test

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2013-01; Primary Completion 2014-09 (Actual); Study Completion 2014-09 (Actual)

PRIMARY OUTCOMES:
Breath carbon monoxide | Throughout study - one year

SECONDARY OUTCOMES:
Saliva cotinine | 2 months, 3 months, 6 months
  When the body processes nicotine, it produces cotinine. Cotinine can be found in saliva.

CONTACTS AND LOCATIONS:
Overall Officials: Jean C. Beckham, Ph.D., Principal Investigator — Duke University Medical Center; VA Medical Center
Locations (1):
- VA Medical Center, Durham, North Carolina, United States

REFERENCES:
- [Derived] Carpenter VL, Hertzberg JS, Kirby AC, Calhoun PS, Moore SD, Dennis MF, Dennis PA, Dedert EA, Hair LP, Beckham JC. Multicomponent smoking cessation treatment including mobile contingency management in homeless veterans. J Clin Psychiatry. 2015 Jul;76(7):959-64. doi: 10.4088/JCP.14m09053. PMID 25699616